CLINICAL TRIAL: NCT02975596
Title: Establishing and Evaluating a School and University Campus-Based Approach to Implementing Serogroup B Meningococcal (MenB) Disease Recommendations in Older Adolescents and Young Adults.
Brief Title: MenB Vaccine: Implementation Via Information, Empowerment and Accessibility
Acronym: MenBVaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201601894; 27449113 (Other Grant/Funding Number: Pfizer, Inc.); IRB201703013 (Other: UF IRB)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Meningococcal Vaccine
Keywords: educational intervention
MeSH Terms: interventions — Immunization Programs; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Youth (Other): Youth between the ages beteen ages 13-18 will be offered awareness, education, empowerment and accessibility intervention components.
  Interventions: Other: Awareness; Other: Education; Other: Empowerment; Other: Accessibility
- College (Other): Age between 18-23 will be offered awareness, education, empowerment and accessibility intervention components.
  Interventions: Other: Awareness; Other: Education; Other: Empowerment; Other: Accessibility
- Adult (Other): parents of adolescents and young adults will be offered awareness, education, and accessibility intervention components.
  Interventions: Other: Awareness; Other: Education; Other: Accessibility
- Parent focus group (No Intervention): Parents discussed barriers and reviewed MenB education materials.
- Provider focus groups (No Intervention): Providers discussed barriers and reviewed MenB education materials.

INTERVENTIONS:
Other: Awareness — Awareness: Conduct an awareness campaign throughout Alachua County to alert the community in general to the significance of Serogroup B meningococcal disease in the United States. To inform the material included in the awareness campaign and the education materials, semi-structured interviews with members for each of the key stakeholder groups: students, parents, and medical practitioners will be conducted.
  Arms: Adult; College; Youth
Other: Education — Education: This component will be both web-based and in-person to meet the individual needs of the learners. There will be parent and a student (18-23 years old) version of the educational curriculum. National resources of patient -focused materials and guidelines will be adapted. There will be pre- and post-education surveys to assess knowledge and vaccine decision-making.
  Arms: Adult; College; Youth
Other: Empowerment — Empowerment: A guided program for adolescents and young adults on "Decision-Making for your Health" will be offered on the vaccination days to assist youth in assessing and utilizing health information to guide their personal decision-making for vaccines.
  Arms: College; Youth
Other: Accessibility — Accessibility: MenB vaccine will be offer on the high school and university campuses through a collaborative program between the local schools, university and department of health. We will offer students booster shots of Men ACWY and HPV at the same time. All vaccines will be offered free of charge. Each vaccine administered will be recorded in Florida SHOTS.
  Arms: Adult; College; Youth

SUMMARY:
As part of an effort to increase MenB vaccine uptake among adolescents and young adults, study teams will conduct qualitative research to maximize the effectiveness of nationally recommended MenB educational materials. In this study, Study Teams will assess local barriers to MenB vaccination by conducting focus groups with parents, students, and health care professionals.

DETAILED DESCRIPTION:
Participants (parents of 16-23 year old teens and young adults, high school and college students 16-23 years old, and health care professionals for 16-23 year olds) will be asked to share their thoughts on the completeness of nationally recommended and publicly available MenB vaccine educational materials in addressing hesitations to receipt of the MenB vaccine. There is no risk in discussing reactions to educational materials. The biggest risk is disclosure of information provided in the study which will be reactions to health-promotion material.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide informed consent or assent

Exclusion Criteria:

* Inability to provide informed consent or assent

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1326 (Actual)
Dates: Start 2016-12; Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Vaccine uptake in adolescents and young adults | 12 months
  Percentage receiving MenB vaccine
Knowledge about MenB vaccine efficacy, potential benefits, possible side effects | 12 months
  Percent of parents and young adults with Men B knowledge

SECONDARY OUTCOMES:
Attitudes re: Meningococcal B vaccine | 12 months
  Pre- and Post- intervention surveys to assess attitudes, perceptions and decision-making re vaccine acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ryan, MD, Principal Investigator — University of Florida
Locations (6):
- United States (6):
  - UF Health Family Medicine and Pediatrics - Magnolia Parke, Gainesville, Florida
  - UF Health Pediatric After Hours, Gainesville, Florida
  - UF Health Pediatrics - Gerold L. Schiebler CMS Center, Gainesville, Florida
  - UF Health Pediatrics - Tower Square, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - UF Family Medicine - Eastside, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soeters HM, McNamara LA, Whaley M, Wang X, Alexander-Scott N, Kanadanian KV, Kelleher CM, MacNeil J, Martin SW, Raines N, Sears S, Vanner C, Vuong J, Bandy U, Sicard K, Patel M; Centers for Disease Control (CDC). Serogroup B Meningococcal Disease Outbreak and Carriage Evaluation at a College - Rhode Island, 2015. MMWR Morb Mortal Wkly Rep. 2015 Jun 12;64(22):606-7. PMID 26068563
- [Background] MacNeil JR, Rubin L, Folaranmi T, Ortega-Sanchez IR, Patel M, Martin SW. Use of Serogroup B Meningococcal Vaccines in Adolescents and Young Adults: Recommendations of the Advisory Committee on Immunization Practices, 2015. MMWR Morb Mortal Wkly Rep. 2015 Oct 23;64(41):1171-6. doi: 10.15585/mmwr.mm6441a3. PMID 26492381
- [Background] Reagan-Steiner S, Yankey D, Jeyarajah J, Elam-Evans LD, Singleton JA, Curtis CR, MacNeil J, Markowitz LE, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years--United States, 2014. MMWR Morb Mortal Wkly Rep. 2015 Jul 31;64(29):784-92. doi: 10.15585/mmwr.mm6429a3. PMID 26225476
- [Background] Hamborsky J, Kroger A, Wolfe CS. Centers for Disease Control and Prevention. Epidemiology and prevention of vaccine-preventable diseases. 13th ed. Washington D.C. Public Health Foundation; 2015.
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] DiClemente RJ, Salazar LF, Crosby RA. A review of STD/HIV preventive interventions for adolescents: sustaining effects using an ecological approach. J Pediatr Psychol. 2007 Sep;32(8):888-906. doi: 10.1093/jpepsy/jsm056. Epub 2007 Aug 27. PMID 17726032
- [Background] Burrus B, Leeks KD, Sipe TA, Dolina S, Soler R, Elder R, Barrios L, Greenspan A, Fishbein D, Lindegren ML, Achrekar A, Dittus P; Community Preventive Services Task Force. Person-to-person interventions targeted to parents and other caregivers to improve adolescent health: a community guide systematic review. Am J Prev Med. 2012 Mar;42(3):316-26. doi: 10.1016/j.amepre.2011.12.001. PMID 22341170
- [Background] Albert D, Chein J, Steinberg L. Peer Influences on Adolescent Decision Making. Curr Dir Psychol Sci. 2013 Apr;22(2):114-120. doi: 10.1177/0963721412471347. PMID 25544805
- [Background] Corbin J, Strauss A. Basics of qualitative research: Techniques and procedures for developing grounded theory. Sage publications; 2014.
- [Background] Centers for Disease Control and Prevention. Adolescent and adult vaccine quiz. http://www2.cdc.gov/nip/adultimmsched/. Accessed 24 June 2016.
- [Background] Tsai Y, Zhou F, Wortley P, Shefer A, Stokley S. Trends and characteristics of preventive care visits among commercially insured adolescents, 2003-2010. J Pediatr. 2014 Mar;164(3):625-30. doi: 10.1016/j.jpeds.2013.10.042. Epub 2013 Nov 25. PMID 24286572
- [Background] Tran CH, Sugimoto JD, Pulliam JR, Ryan KA, Myers PD, Castleman JB, Doty R, Johnson J, Stringfellow J, Kovacevich N, Brew J, Cheung LL, Caron B, Lipori G, Harle CA, Alexander C, Yang Y, Longini IM Jr, Halloran ME, Morris JG Jr, Small PA Jr. School-located influenza vaccination reduces community risk for influenza and influenza-like illness emergency care visits. PLoS One. 2014 Dec 9;9(12):e114479. doi: 10.1371/journal.pone.0114479. eCollection 2014. PMID 25489850
- [Background] Livingston MD, Komro KA, Wagenaar AC. The effects of survey modality on adolescents' responses to alcohol use items. Alcohol Clin Exp Res. 2015 Apr;39(4):710-5. doi: 10.1111/acer.12659. Epub 2015 Mar 9. PMID 25752744
- [Background] Edwards PJ, Roberts I, Clarke MJ, Diguiseppi C, Wentz R, Kwan I, Cooper R, Felix LM, Pratap S. Methods to increase response to postal and electronic questionnaires. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):MR000008. doi: 10.1002/14651858.MR000008.pub4. PMID 19588449
- [Background] Faes C, Molenberghs G, Aerts M, Verbeke G, Kenward MG. The effective sample size and an alternative small-sample degrees-of-freedom method. Am Stat. 2009 Nov 1;63(4):389-99.
- [Background] Yuan CT, Nembhard IM, Stern AF, Brush JE Jr, Krumholz HM, Bradley EH. Blueprint for the dissemination of evidence-based practices in health care. Issue Brief (Commonw Fund). 2010 May;86:1-16. PMID 20469542
- [Derived] Richardson E, Ryan KA, Lawrence RM, Harle CA, Desai SM, Livingston MD, Rawal A, Staras SAS. Increasing awareness and uptake of the MenB vaccine on a large university campus. Hum Vaccin Immunother. 2021 Sep 2;17(9):3239-3246. doi: 10.1080/21645515.2021.1923347. Epub 2021 Jun 2. PMID 34076556